CLINICAL TRIAL: NCT04891731
Title: Efficacy and Safety of Leuprorelin Acetate Every-3-months Depot Plus an Aromatase Inhibitor or Tamoxifen in Premenopausal Women With Hormone Receptor-positive Breast Cancer: a Clinical Prospective Observational Study
Brief Title: Efficacy and Safety of Leuprorelin 3M in Premenopausal Women With Hormone Receptor-positive Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liu Qiang, Doctor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SunYatsenU2H-LQ5
Record Dates: First submitted 2021-05-17; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Hormone Receptor-positive Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- leuprorelin 3M plus AIs: leuprorelin 3M: 11.25 mg subcutaneous administration every 3 months for 1 year AIs: anastrozole 1mg /letrozole 2.5mg/exemestane 25mg daily for 1 year
  Interventions: Drug: AI or TAM
- leuprorelin 3M plus TAM: leuprorelin 3M: 11.25 mg subcutaneous administration every 3 months for 1 year TAM: daily for 1 year
  Interventions: Drug: AI or TAM

INTERVENTIONS:
Drug: AI or TAM — This is an observational study, the researcher will describe the ratio of E2 control between leuprorelin plus TAM or leuprorelin plus AIs patients based on the actual clinical use.

SUMMARY:
Leuprorelin, a LHRH agonist, acts as a potent inhibitor of gonadotropin secretion and is commonly used for the treatment of hormone-responsive prostate cancer, premenopausal HR+ breast cancer, endometriosis and uterine fibroids. It is currently available in 1M, 3M, 6M for subcutaneous administration. Initially administration would stimulate an increase in LH and FSH, causing a transient increase of E2 in 2-4 weeks. Continuous administration results in a subsequent decrease in E2 levels, as a result of decreased levels of luteinizing LH and FSH. After stopping injection, ovarian function could gradually recover. Adverse events related to leuprorelin include flushing, mood swings and urogenital symptoms.

At present, the treatment of premenopausal breast cancer mainly includes 1M and 3M GnRHa. Leuprorelin 11.25mg dosage form is currently the only 3M GnRHa in China that has gotten breast cancer indications. The use of 3M GnRHa could improve patients' compliance and reduce injection discomfort. However, previous studies about GnRHa alone or in combination with TAM or AIs usually used 1M GnRHa. There have been few studies reporting the suppression effects of E2 levels and clinical outcome with leuprorelin 3M in combination with TAM or AIs.

DETAILED DESCRIPTION:
Background:

There are some differences in the age of onset of breast cancer, histopathological types, and treatment methods between Asians and non-Asians. Incidence peaks at age 40-50 in Asian women, with more than half of premenopausal patients, but 65-70 years in US women, most of which are postmenopausal[1]. Besides, compared with Americans, Asian women younger than 50 have a higher prevalence of luminal A breast cancer and less basal-like subtype. Therefore, the application of OFS has always been the focus for the treatment of premenopausal women with HR+ breast cancer in Asia.

OFS therapy includes oophorectomy, ovarian radiation, and the use of GnRHa. Several studies have shown that the use of GnRHa in premenopausal women can achieve similar efficacy to oophorectomy and ovarian radiation therapy. As GnRHa has the advantages of non-invasiveness and reversibility, it has gradually replaced oophorectomy and ovarian radiation, and has become the main method of OFS in premenopausal women with HR+ breast cancer. Meanwhile, GnRHa in combination with TAM or AIs is increasingly used for premenopausal HR+ breast cancer patients. Previous studies have revealed that GnRHa alone or in combination with TAM or AIs has shown effective estrogen suppression and certain survival benefits for most patients with breast cancer. In addition, the 5-year follow-up results of the TEXT / SOFT study in 2014 showed that compared with OFS + TAM, OFS + AI treatment significantly improved DFS, prolonged cancer-free survival time and distant recurrence-free metastasis[8, 9]. The 9-year follow-up results of the TEXT / SOFT study in 2019 indicated that OFS + AI versus OFS + TAM or TAM single drugs, years of distant recurrence risk in patients with high risk of recurrence have an absolute benefit rate of 10-15 %, Intermediate risk is 4-5%, low-risk benefit is not obvious. In 2019, the ABCCG reviewed ESO-ESMO and St. Gallen's treatment recommendations for HR+/ Her-2 negative breast cancer in premenopausal women, discussed controversial issues and pointed out that patients with low recurrence risk can be treated with TAM alone. For patients with high risk of recurrence, chemotherapy + OFS + AI should be given. It indicates that not all premenopausal HR+ patients with early breast cancer need auxiliary OFS, and more clinical trials on OFSin premenopausal HR + patients are necessary and worthwhile.

Leuprorelin, a LHRH agonist, acts as a potent inhibitor of gonadotropin secretion and is commonly used for the treatment of hormone-responsive prostate cancer, premenopausal HR+ breast cancer, endometriosis and uterine fibroids. It is currently available in 1M, 3M, 6M for subcutaneous administration. Initially administration would stimulate an increase in LH and FSH, causing a transient increase of E2 in 2-4 weeks. Continuous administration results in a subsequent decrease in E2 levels, as a result of decreased levels of luteinizing LH and FSH. After stopping injection, ovarian function could gradually recover. Adverse events related to leuprorelin include flushing, mood swings and urogenital symptoms.

At present, the treatment of premenopausal breast cancer mainly includes 1M and 3M GnRHa. Leuprorelin 11.25mg dosage form is currently the only 3M GnRHa in China that has gotten breast cancer indications. The use of 3M GnRHa could improve patients' compliance and reduce injection discomfort. However, previous studies about GnRHa alone or in combination with TAM or AIs usually used 1M GnRHa. There have been few studies reporting the suppression effects of E2 levels and clinical outcome with leuprorelin 3M in combination with TAM or AIs.

To further investigate the suppression effects of E2 levels of 3M GnRHa, we conducted a single-arm, prospective clinical observational study evaluating the efficacy and safety of adjuvant therapy with leuprorelin 3M in combination with TAM or AIs in premenopausal HR+ breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. age≥18 years;
2. Tumor that expressed ER or progesterone receptor in at least 10% of the cells, as assessed by immunohistochemical testing
3. T1 to T3, any N, and M0, according to the TNM classification
4. Any type of breast surgical procedure
5. Any type of preoperative and/or postoperative adjuvant chemotherapy prior to enrollment
6. Capable of receiving the study drug within 12 weeks after surgery or after postoperative chemotherapy completion prior to enrollment
7. Eastern Cooperative Oncology Group performance status of Grade 0 or 1

Exclusion Criteria:

1. Bilateral oophorectomy or ovarian irradiation
2. No use of other OFS drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Premenopausal patients with histologically confirmed hormone receptor-positive breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
the suppression proportion of serum estradiol (E2) | March,2023
  The suppression proportion of serum estradiol (E2) to the menopausal level (E2≤30 pg/mL) at different time points (4, 12, 24, 36 and 48 weeks) during the first year for leuprorelin 3M depot plus TAM or AIs.

SECONDARY OUTCOMES:
Quality of Life (QoL) | March,2023
  To evaluate the Quality of Life (QoL) of Patient who receive Leu 3M depot for OFS treatment evaluated by FACT-B and FACT-ES questionnaire.
Adverse events(AEs) | March,2023
  To observe the incidence of adverse events(AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Liu, MD, Principal Investigator — Sunyat-sen Memorial Hospital

IPD SHARING:
Plan to Share IPD: Undecided